CLINICAL TRIAL: NCT03131700
Title: Phase I, Double Blind, Randomized, Parallel-Arm, Single-Dose, Bioequivalence and Safety Study of Bevacizumab-biosimilar (RPH-001) Compared to Bevacizumab-innovator (Avastin®, Roche) in Healthy Male Volunteers
Brief Title: Bioequivalence and Safety Study of Bevacizumab-biosimilar (RPH-001) Compared to Bevacizumab-innovator
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision of the Sponsor
Sponsor: TRPHARM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RPH001BEV01
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: RPH101; RPH-101; Biosimilar; Bevacizumab; Safety
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-001 (Experimental): A single dose of RPH-001 will be administered (IV) 5 mg/kg dose .
  Interventions: Biological: RPH001
- EU sourced Avastin® (Active Comparator): A single dose of Avastin® will be administered (IV) 5 mg/kg dose .
  Interventions: Biological: Avastin®

INTERVENTIONS:
Biological: RPH001 — Avastin® has been approved for treatment of various cancers in many countries of the world including the USA, EU countries, and Turkey. In Turkey, Avastin® is approved with a different trade name, Altuzan®, for treatment of metastatic colorectal cancer.
  Arms: RPH-001
Biological: Avastin® — R-Pharm created a biological analog of Avastin®, RPH-001. RPH-001 and Avastin® have similar physicochemical properties, pharmacokinetic profile and affinity to human vascular endothelial growth factor, similar toxicity and efficacy confirmed by preclinical study results.
  Other Names: Bevacizumab
  Arms: EU sourced Avastin®

SUMMARY:
The purpose of this to assess pharmacokinetic bioequivalence between two bevacizumab products, RPH-001 (TRPHARM) and EU sourced Avastin® (Roche), after single IV administration at 5 mg/kg fixed dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 55 years inclusive.
* Adult healthy male subjects between 18.0 and 30.0 kg/m2 body mass index (inclusive) and body weight ≥ 60 kg and ≤ 100 kg (inclusive).

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol test at screening or baseline visits

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration | Until 100 days after administration
  Cmax
Area under concentration-time curve from time zero to the last sampling time | Until 100 days after administration
  Area Under the Curve - AUC(0-t)
Area under concentration-time curve from time zero to infinity | Until 100 days after administration
  Area Under the Curve - AUC(0-∞)

SECONDARY OUTCOMES:
Concentration-time profiles | Until 100 days after administration
  RPH-001 and Avastin®
Time to maximum concentration (Tmax) | Until 100 days after administration
  RPH-001 and Avastin®
Terminal elimination half-life (t½) | Until 100 days after administration
  RPH-001 and Avastin®
Terminal elimination rate constant (λz) | Until 100 days after administration
  RPH-001 and Avastin®
Apparent volume of distribution (Vz) | Until 100 days after administration
  RPH-001 and Avastin®
Clearance (CL) | Until 100 days after administration
Volume of distribution at steady state (Vss) | Until 100 days after administration
Nature, frequency, severity and relationship to study drug of recorded adverse events | Until 100 days after administration
Physical examination | Until 100 days after administration
Heart rate | Until 100 days after administration
Blood Pressure | Until 100 days after administration
Respiratory rate | Until 100 days after administration
Oxygen saturation | Until 100 days after administration
Body temperature | Until 100 days after administration
ECG | Until 100 days after administration
Clinical laboratory tests | Until 100 days after administration
Anti-drug-antibody (ADA) | Until 100 days after administration
Neutralizing antibody (NAb) | Until 100 days after administration

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Sezer, PHD, Principal Investigator — IKUM